CLINICAL TRIAL: NCT06821074
Title: Comparative Study of Visual Function Training With Defocus-Enhanced Spectacles vs. Single Vision Spectacles on Myopia Control in Children
Brief Title: Defocus-Enhanced vs. Single Vision Spectacles in Myopia Control Visual Function Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Visionly Plus Eye Hospital (Other)
Collaborators: High Myopia Control Alliance (HIMALAYA) (Unknown); Beijing New Vision Eye Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Himalaya202502
Record Dates: First submitted 2025-02-10; First posted 2025-02-11 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Myopia
Keywords: myopia; Visual Function Training; Defocus-Enhanced Spectacles; Single Vision Spectacles
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Defocus-enhanced spectacles (Experimental): Vision function training while wearing defocus-enhanced spectacles
- Single vision spectacles (Placebo Comparator): Vision function training while wearing single vision spectacles
  Interventions: Device: Single vision spectacles

INTERVENTIONS:
Device: Defocus-enhanced spectacles — Vision function training while wearing defocus-enhanced spectacles
Device: Single vision spectacles — Vision function training while wearing single vision spectacles
  Arms: Single vision spectacles

SUMMARY:
The purpose of this study is to compare the effectiveness of vision function training using defocus-enhanced spectacles (DIMS) versus single vision spectacles combined with vision function training in controlling myopia progression in children aged 6-18 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-18 years.
* Diagnosed myopia with SER between -0.50D and -4.00D.
* Astigmatism ≤ 2.50DC.
* Anisometropia < 1.25D.

Exclusion Criteria:

* Suspected genetic syndromes (e.g., Stickler, Marfan).
* Other eye diseases (e.g., glaucoma, cataracts, retinal abnormalities, strabismus).
* Myopia progression <0.50D SER in the last year.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in spherical equivalent 12 months after the commencement of training. | Regular sessions commenced from the day of the initial training and continued until 12 months after the first visual training session.
  Change in spherical equivalent 12 months after the commencement of training.

SECONDARY OUTCOMES:
Change in axial length 12 months after the commencement of training. | Regular sessions commenced from the day of the initial training and continued until 12 months after the first visual training session.
  Change in axial length 12 months after the commencement of training.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing New Vision Eye Hospital, Beijing
  - Beijing Visionly Plus Eye Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: February 2025-February 2027